CLINICAL TRIAL: NCT00825136
Title: A Study on Mental Health Care by Using Specific Vital Signs
Brief Title: Treatment of Panic Disorder Via Internet With a Wireless Temperature Biofeedback Ring
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The main limitations were the small sample size and low completion rate.
Sponsor: Chimei Medical Center (Other)
Responsible Party: Principal Investigator, Fong-Lin Jang, Department of Psychiatry, Chimei Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 09707-001
Record Dates: First submitted 2009-01-15; First posted 2009-01-19 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Panic Disorder
Keywords: Panic Disorder; Temperature Biofeedback; Internet
MeSH Terms: conditions — Panic Disorder | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- relaxation (Active Comparator): The patients of this arm practice on-line muscle relaxation for 8 weeks.
  Interventions: Behavioral: relaxation
- relaxation & biofeedback (Experimental): The patients of this arm practice on-line muscle relaxation plus finger temperature biofeedback for 8 weeks.
  Interventions: Behavioral: relaxation; Behavioral: biofeedback (finger temperature biofeedback)

INTERVENTIONS:
Behavioral: relaxation — Participants were asked to log in the system to keep the muscle relaxation program every day and complete some self-rating scales on browser every week.
Behavioral: biofeedback (finger temperature biofeedback) — Participants were asked to log in the system to keep the muscle relaxation program plus finger temperature biofeedback every day and complete some self-rating scales on browser every week.
  Arms: relaxation & biofeedback

SUMMARY:
Internet plays a more and more important role in many applications of healthcare. Many researches on the integrations of internet and mental health care have been proposed in recent years. This project aims at the development of an online treatment system which combines the biofeedback therapy and the web technologies to treat the patients suffering from panic disorder with partial response to medications. This project also evaluates the efficacy of a new- designed wireless temperature biofeedback ring.

DETAILED DESCRIPTION:
The participants should be chronic panic patients. They login an web-based server and practice muscle relaxation on-line every day. There will be two two parallel groups: one group practicing muscle relaxation only and the other practicing muscle relaxation with finger surface temperature monitor through a wireless biofeedback ring.

ELIGIBILITY:
Inclusion Criteria:

1. The participant must fulfill DSM-IV criteria for panic disorder.
2. The participant must be between 18 and 60 years of age.
3. The participant must have panic disorder as the primary problem.
4. If the participant is taking prescribed drugs for panic disorder, a) the dosage have to be constant for 2 months before starting treatment, and b) the participant have to agree to keep the dosage constant for 1 month after starting treatment.
5. If the participant was already in therapy, the contact must have lasted at least 6 months and not be based on cognitive behavior therapy.
6. All participants have access to a computer with an Internet connection.

Exclusion Criteria:

1. The participant suffers from any other psychiatric disorder in immediate need of treatment.
2. The participant fulfills DSM-IV criteria for major depression.
3. The participant has epilepsy, kidney problems, strokes, organic brain syndrome, emphysema, heart disorders, or chronic hypertension. 4. The participant has alcoholism.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
score change of The Panic Disorder Severity Scale(PDSS) | day 1 / 4 weeks/ 8 weeks

SECONDARY OUTCOMES:
score change of MOS 36-Item Short-Form Health Survey (SF-36) | day 1 / 4 weeks/ 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fong-Lin Jang, M.D., Study Director — Chimei Medical Center
Locations (1):
- Psychiatry Department, Chimei Medical Center, Tainan, Taiwan